CLINICAL TRIAL: NCT01958996
Title: Phase I/II Study of Escalating Doses of Idarubicin Orally Given With Oral Cyclophosphamide, Etoposide, Prednisolone and Intravenous Rituximab in Elderly Patient With Disseminated High Grade Non Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: OROCIEP
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: High Grade Lymphomas CD20 Positive
MeSH Terms: interventions — Idarubicin

ARMS (1):
- idarubicin (Experimental)
  Interventions: Drug: idarubicin

INTERVENTIONS:
Drug: idarubicin

SUMMARY:
R-CHOP with doxorubicin is the standard first line treatment of high grade non-Hodgkin's lymphoma. In order to avoid central venous system insertion and reduce hospitalization time in elderly patients, we developed an oral chemotherapy treatment: " OROCIEP"trial.

Nineteen patients were enrolled and 127 chemotherapy cycles were available for toxicities. The estimated two-years overall survival was 74%. The main haematological toxicity was neutropenia.

This study is still ongoing to confirm recommended dose of oral anthracycline.

ELIGIBILITY:
Inclusion Criteria:

* CD20-positive diffuse large B-cell lymphoma.WHO classification (55)
* Written informed consent
* Age > 65 and < 80 years
* Performance status (ECOG) <3
* measurable disease
* Serology HIV negative, Hepatites B, Hepatites C negative

Exclusion Criteria:

* Serology HIV positive, Hepatite B positive, Hepatite C positive
* Cardiac failure.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2009-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of idarubicin | 9 months

SECONDARY OUTCOMES:
Remission rate after 4 cycles and 8 cycles | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

REFERENCES:
- [Derived] Guidez S, Lacotte-Thierry L, Tomowiak C, Princet I, Dreyfus B, Olivier G, Fleck E, Corby A, Motard C, Barrier J, Machet A, Le Du K, Debiais-Delpech C, Chabin M, Leleu X, Guilhot J, Delwail V. Oral CHOP-like chemotherapy in 60-80 years-old patients with diffuse large B-cell lymphoma. Br J Haematol. 2019 Sep;186(6):e175-e178. doi: 10.1111/bjh.16056. Epub 2019 Jul 15. No abstract available. PMID 31309541